CLINICAL TRIAL: NCT01948726
Title: Multicenter Phase-II-Trial of Evaluation of Acute Toxicity in Hypofractionation With Simultaneous Integrated Boost for Early Breast Cancer
Brief Title: Hypofractionation With Simultaneous Integrated Boost for Early Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Schleswig-Holstein (Other)
Collaborators: University of Luebeck (Other)
Responsible Party: Principal Investigator, Juergen Dunst, Prof., Prof. Dr. med. Juergen Dunst, University Hospital Schleswig-Holstein
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARO 2013-04
Record Dates: First submitted 2013-08-23; First posted 2013-09-24 (Estimated); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Breast Cancer After Breast Conserving Surgery Indicating Postoperative Radiotherapy With Boost
Keywords: Breast cancer; Hypofractionation; Simultaneous integrated boost; Toxicity
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hypofractionation with SIB (Experimental)
  Interventions: Radiation: Hypofractionation with simultaneous integrated boost

INTERVENTIONS:
Radiation: Hypofractionation with simultaneous integrated boost

SUMMARY:
Hypofractionation with simultaneous integrated boost has been investigated in a few trials and appears to be safe and feasible with less lung toxicity in smaller studies.

Investigators initiated this multicenter phase II prospective trial to analyse acute toxicity of hypofractionation with simultaneous integrated boost in patients with early breast cancer under the hypothesis that the ratio of patients with acute radiogenic toxicity Grad II according NCI-CTCAE amounts maximum 20%.

DETAILED DESCRIPTION:
Hypofractionated radiotherapy of the breast 16 × 2.50 Gy with simultaneous integrated boost to the tumor bed (total dose within the boost volume 16 × 3.00 Gy).

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically confirmed breast cancer operated by breast conserving surgery with clear margins
* Indication to adjuvant radiotherapy including boost radiotherapy
* Clearly identified primary tumor region preferably by radiopaque clips
* Primary wound healing after breast conserving therapy without signs of infection
* Pre- and/or postoperative chemotherapy and endocrine therapy were permitted when indicated
* Written informed consent

Exclusion Criteria:

* Patients operated by mastectomy
* No indication for boost radiation
* Resection margins positive for disease or insufficient identification of the boost volume
* Indication for radiotherapy of the regional lymph nodes
* History of prior breast or thoracic radiotherapy
* Extended postoperative seroma at the beginning of radiotherapy
* Psychiatric disorders or psychological disabilities thought to adversely affect treatment compliance
* Pregnant or lactating patients and woman of child bearing potential, who lacked effective contraception

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2013-12; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Acute Skin Toxicity | 6 months
  Acute skin radiogenic toxicity grade II or higher according to NCI-CTCAE

SECONDARY OUTCOMES:
Number of Patients treated on Protocol | 22-29 days (16 fractions)
  Dose constraints Dmedian lung < 10 Gy; Dmedian heart < 5 Gy, Dmax ≤ 40 Gy; Dmedian anterior branch of the left coronary artery (LAD, RIVA) < 15 Gy, Dmax ≤ 40 Gy; Dmedian contralateral breast < 3 Gy
Acute General Toxicity | 0 to 6 months
  All dimensions of NCI-CTCAE
Quality of life Score | 0 to 6 months
  EORTC QLQ-C30, -BR23
Performance | 0 to 6 months
  ECOG

OTHER OUTCOMES:
Skin toxicity (Cosmetic results) | 0 to 6 months
  NCI-CTCAE

CONTACTS AND LOCATIONS:
Overall Officials: Juergen Dunst, Prof., Study Chair — University Medical Center Schleswig-Holstein (UKSH)
Locations (19):
- Germany (19):
  - Charité University Medical Center Berlin, Berlin
  - Krankenhaus Buchholz, Buchholz
  - Klinikum des Landkreises Deggendorf Mammazentrum, Deggendorf
  - Praxis für Strahlentherapie am Krankenhaus Dresden-Friedrichstadt, Dresden
  - Malteser St. Franziskus-Hospital, Flensburg
  - Onkologischer Schwerpunkt (OSP) Goeppingen, Göppingen
  - Strahlenzentrum Hamburg Nord, Hamburg
  - Radiologie and Radioonkologie, Hamburg
  - University Medical Center Schleswig-Holstein (UKSH), Department of Radiotherapy, Campus Kiel, Kiel
  - University Medical Center Schleswig-Holstein (UKSH), Department of Radiotherapy, Campus Luebeck, Lübeck
  - MGZ Luebeck im Hochschulstadtteil, Lübeck
  - Staedtisches Klinikum Lueneburg, Lüneburg
  - University Medical Center Mainz, Department of Radiotherapy, Mainz
  - University Medical Center Rechts der Isar Department of Radiotherapy Muenchen, München
  - Radiology Pinneberg, Pinneberg
  - Helios Kliniken Schwerin, Schwerin
  - Johanniter-Krankenhaus Genthin-Stendal, Stendal
  - MVZ Klinikum Straubing GmbH, Straubing
  - Heinrich-Braun-Klinikum Zwickau, Zwickau